CLINICAL TRIAL: NCT02461849
Title: A Phase II, Open-label, Study in Patients With Refractory, Metastatic Cancer Harboring KIT Mutation or Amplification to Investigate the Clinical Efficacy and Safety of Imatinib Therapy
Brief Title: Patients With Refractory, Metastatic Cancer Harboring KIT Mutation or Amplification to Investigate the Clinical Efficacy and Safety of Imatinib Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-12-074
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Advanced, Refractory Cancer
MeSH Terms: conditions — Neoplasms | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib (Experimental): Imatinib 400mg qd daily Until disease progression, patient's refusal
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Imatinib 400mg qd daily

SUMMARY:
KIT is a receptor tyrosine kinase that binds to stem-cell factor (SCF), activating a series of downstream effector pathways. KIT is an established therapeutic target in cancer with activating mutations of KIT, such as gastrointestinal stromal tumors (GIST), and significant benefit is achieved with various small molecule inhibitors of KIT such as imatinib mesylate. Moreover, there is increasing evidence implicating KIT mutations as tractable therapeutic targets in melanoma. Additional information is required to characterize the functional role of low-frequency mutations in KIT and to determine whether amplification of wild type KIT is a real driver that can be targeted therapeutically. Except GIST and melanoma, other solid cancers were reported to have KIT mutation even in low frequency. A molecular profiling of the tumors of patients referred to the phase I clinic at the M.D. Anderson Cancer Center showed KIT mutation in 7 patients in total of 431 patients (2%).

Hence, the investigators planned this study to apply the molecularly targeted agent, imatinib to various types of cancers harboring KIT mutation or amplification.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 20
2. advanced, refractory cancer patients who failed standard of care (SOC)
3. KIT aberration: defined as mutation in exons 9, 11, 13, 17 or 18, or nanostring CNV by quantitative PCR (greater than 3 copies) or subject with specific sensitivity (Z-score<-1) to imatinib by Avatar scan whose disease has progressed following standard therapy or that has not responded to standard therapy or for which there is no standard therapy
4. ECOG performance status of 0~2
5. measurable or evaluable lesion per RECIST 1.1 criteria
6. adequate marrow, hepatic, renal and cardiac functions

   * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN), or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy
   * Total serum bilirubin ≤ 1.5 x ULN
   * Absolute neutrophil count(ANC) ≥ 1,500/uL
   * Platelets ≥ 100,0000/uL
   * Hemoglobin ≥ 9.0 g/dL
7. provision of a signed written informed consent

Exclusion Criteria:

1. severe co-morbid illness and/or active infections
2. pregnant or lactating women
3. history of major surgery or radiotherapy within 4 weeks
4. active CNS metastases not controllable with radiotherapy or corticosteroids (however, CNS metastases (except for leptomeningeal seeding) are allowed if controlled by gamma knife surgery or surgery or radiotherapy or steroid)
5. known history of hypersensitivity to study drugs

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04-04 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | expected average of 24 weeks
  Response will be evaluated according to RECIST(Response Evaluation Criteria In Solid Tumors) 1.1 guidelines.Tumor responses will be assessed after the 2cycle chemotherapy and after completion of treatment. They should be classified as complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD) according to the Revised Response Criteria for refractory, metastatic cancer harboring KIT mutation or amplification.

SECONDARY OUTCOMES:
Duration of response | expected average of 24 weeks
Progression-free survival | expected average of 24 weeks
Overall survival | expected average of 3years
Number of subjects with Adverse Events as a measure of safety | expected average of 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea